CLINICAL TRIAL: NCT02810262
Title: Association of Bone and Metabolic Parameters With Overall Survival in Patients With Bone Metastases From Adenocarcinoma Lung Cancer (POUMOS)
Acronym: POUMOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50772
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Bone Metastases; Lung Cancer
Keywords: Lung cancer; Bone metastases; EGFR; KRAS; Bone biomarkers; Metabolic parameters
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine Serum and plasma Bone biopsy Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- First bone metastasis of adenocarcinoma lung cancer: Patients entering the group have a suspected first bone metastasis of adenocarcinoma lung cancer and should undergo bone biopsy to histologically prove the diagnosis.
  Interventions: Other: Bone metastases biopsy

INTERVENTIONS:
Other: Bone metastases biopsy — The vast majority of bone biopsy are performed under CT-scan. In some rare cases, the histology will be performed during surgery (either biopsy of the bone metastasis or surgical piece when treating a fracture).

SUMMARY:
Mortality due to non small cell lung cancers is the first cause of cancer death in men around the world. Lung adenocarcinoma regularly induces bone metastases responsible for high morbidity and impaired life quality. Overall survival of these patients is poor. Thus the investigators aimed to identify if some bone and metabolic parameters were associated with overall survival.

Patients and Methods POUMOS is a prospective cohort of patients suffering from adenocarcinoma lung cancers with a first bone metastasis (stage IV). All patients have a bone biopsy with molecular status characterization of the tumor for EGFR, KRAS, BRAF and ALK. Bone metastasis localizations are obtained by bone scintigraphy or FDG-PET/CT. Whole body composition is obtained by DEXA scan (Hologic®). The investigators assessed also fasting blood levels of bone and metabolic biomarkers.

Survival analyses will be performed using a proportional hazard regression model.

ELIGIBILITY:
Inclusion Criteria:

* adults over 18 years
* both gender
* covered by the French National Insurance
* first bone metastases of adenocarcinoma lung cancer (synchronous or metachrone)

Exclusion Criteria:

- adenocarcinoma previously treated by systemic oncologic treatment (chemotherapy, targeted therapy, immunotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: POUMOS is a prospective cohort of patients suffering from adenocarcinoma lung cancers with a first bone metastasis (stage IV). All patients have a bone biopsy with molecular status characterization of the tumor
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-06; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
serum DKK1 | day 0
  Biomarkers are assessed at baseline.

SECONDARY OUTCOMES:
serum HbA1C | day 0
  Biomarkers are assessed at baseline
urinary CTX | day 0
  Biomarkers are assessed at baseline
hip bone mass (g/cm²) | day 0
  Whole body densitometry is performed at baseline
mutational profile of the bone metastases | day 0
  Molecular characterization of the bone metastases by PCR (EGFR, KRAS, BRAF) and FISH (ALK)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hôpital Edouard Herriot - Centre des Métastases Osseuses (CEMOS), Lyon, France

REFERENCES:
- [Derived] Dirckx N, Tower RJ, Mercken EM, Vangoitsenhoven R, Moreau-Triby C, Breugelmans T, Nefyodova E, Cardoen R, Mathieu C, Van der Schueren B, Confavreux CB, Clemens TL, Maes C. Vhl deletion in osteoblasts boosts cellular glycolysis and improves global glucose metabolism. J Clin Invest. 2018 Mar 1;128(3):1087-1105. doi: 10.1172/JCI97794. Epub 2018 Feb 12. PMID 29431735